CLINICAL TRIAL: NCT06452368
Title: Palatal Versus Buccal Protraction Using Plates Assisted With Facemask in Growing Class III Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Mohamed Adel Raghib, Phd researcher, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M04020822
Record Dates: First submitted 2024-06-05; First posted 2024-06-11 (Actual); Last update posted 2024-06-14 (Actual); Status verified 2024-06

CONDITIONS: Class III Malocclusion
MeSH Terms: conditions — Malocclusion, Angle Class III

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Palatal protraction (Active Comparator): Palatal plate assisted with facemask
  Interventions: Device: facemask
- Buccal protraction (Active Comparator): Buccal plate assisted with facemask
  Interventions: Device: facemask

INTERVENTIONS:
Device: facemask — Fixation of miniplates by four screws in the maxilla and protraction by using facemask

SUMMARY:
to compare Palatal and buccal protraction using plates assisted with facemask in growing class III patients

DETAILED DESCRIPTION:
A randomized controlled clinical trial was adopted in this study. A total of 20 growing Class III patients were selected from patients seeking orthodontic treatment. The participants were recruited from the department of Orthodontics at Faculty of Dentistry, Mansoura University. No active advertisement was used for participant recruitment, and instead, a convenience sample was formed. Prior to participating in the study, the purpose of the study was explained to the parents of the children and informed consents and assents were obtained according to the guidelines on human research adopted by the Research Ethics Committee Faculty of Dentistry, Mansoura University

ELIGIBILITY:
Inclusion Criteria:

* Growing patients with age ranged between 8-13 years old.
* Patients should have examination: Class III malocclusion due to maxillary retrusion as verified by clinical and radiographic examination; SNA <79 and ANB angle < -1.
* Good likelihood of recall availability.

Exclusion Criteria:

* Vertical skeletal mal relationship.
* History of previous orthodontic/orthopedic treatment.
* Bad habits that may jeopardize the appliance.
* Patients with systemic diseases
* Congenital deformities such as cleft lip and/or palate.

Ages: 8 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2023-11-20 (Actual)

PRIMARY OUTCOMES:
cephalometric radiographs | 12 month
  cephalometric radiographs were analyzed and the amount of maxillary protraction, the dentoskeletal as well the soft tissue changes were evaluated

CONTACTS AND LOCATIONS:
Locations (1):
- Mohamed Adel Raghib, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No